CLINICAL TRIAL: NCT02461277
Title: Postoperatory Recovery in Thoracic Surgical Procedure, Fast-track Protocol vs. Conventional Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Sâmia Geórgia Dantas Linhares, Physiotherapist, Instituto do Coracao
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Heart Institute InCor
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Thoracic Surgery
Keywords: postoperative care; exercise test; early ambulation; Fast-track

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fast-track protocol (Active Comparator): Before surgery, patients are informed about the surgical procedure, anesthesia and rehabilitation protocol. The surgery occurs in accordance with the principles of the Fast-track: minimal invasive surgery, epidural anesthetic management, avoiding the need opioid in postoperatory analgesia and use of an standardized postoperatory management protocol to an early oral intake and early mobilization.
  Interventions: Other: Fast-track protocol
- Conventional care (No Intervention): Usual care routine postoperative

INTERVENTIONS:
Other: Fast-track protocol — Preoperatory management, epidural anesthetic management, avoiding the need opioid in postoperatory analgesia and use of an standardized postoperatory management protocol to an early oral intake and early mobilization. At the postoperative recovery room, after extubation and fully awake, patients started physiotherapy exercises, as physical exercises of moving up upper and lower extremities accompanied by deep breathing exercises. After than, the patients standed up beside the bed and if there was no complications, patients performed ambulation. The physiotherapist aided the patients during all period.
  Other Names: Early rehabilitation
  Arms: Fast-track protocol

SUMMARY:
The aim of this study was to compare the functional capacity of exercise by six-minute walk test before and after thoracic surgical procedure in subjects who have undergone the Fast-track protocol with those who were under conventional care. Researchers want to find out if Fast-track is a strategy to enhance functional capacity after thoracic surgery.

DETAILED DESCRIPTION:
Fast track programs represents a new approach to the management of patients undergoing surgery. It is perioperative care pathway designed to achieve early recovery and helps to minimize postoperative morbidity and mortality.

These multimodal approaches focuses on enhancing recovery and reducing of surgical stress by minimal invasive surgery, optimized pain relief, early nutrition and ambulation.

In postoperative, the bed rest leads to the increase in muscle loss and weakness, impairs pulmonary function, predisposes to venous stasis and thromboembolism, increases infection complications and reduces functional capacity.

However, information on the results of Fast-track protocols in functional capacity of exercise during hospital stay is sparse.

The six-minute walk test is use to measure of functional capacity of exercise in different populations and to detect changes after interventions. The distances traveled in two six-minute walk test (preoperative and postoperative) will be compared between the two groups (Fast-track and Conventional).

In this trial the investigators will consider Fast-track protocol to be feasible to enhance functional capacity of exercise after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo a thoracic surgical procedure
* sign the informed consent form
* independent ambulation
* ability to understand and follow instructions

Exclusion Criteria:

* contraindications for epidural catheter placement
* refusal to do physical exercises on postoperative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Functional capacity of exercise ( six-minute walk test) | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Change from baseline in distance walking on hospital discharge

SECONDARY OUTCOMES:
Time to first postoperative ambulation | up 2 hour after surgery
  Time from end of surgical procedure until first postoperative ambulation
The length of hospital stay | expected average of 6 days
  Time to achieve standardized hospital discharge criteria (tolerance of oral intake, recovery of lower gastrointestinal function, adequate pain control on oral analgesia, ability to mobilize and self care and no evidence of complications or untreated medical problems).
Surgical complications | up 6 days after surgery
  Pneumonia, atelectasis, pneumothorax and air leak in the chest drainage